CLINICAL TRIAL: NCT01972776
Title: A Two Part, Double Blind, Placebo Controlled, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Multiple Doses of QBM076 in Patients With COPD
Brief Title: A Safety, Tolerability and Efficacy Study in Chronic Obstructive Pulmonary Disease (COPD) Patients With QBM076.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Part 1 was completed. Part 2 was terminated for safety reasons.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CQBM076X2203; 2012-005615-92 (EudraCT Number)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: COPD
Keywords: COPD, inflammation, small airways, LCI, PFTs, lung heterogeneity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- QBM076 Part 1 Cohort 1 (Experimental): Participants received QBM076 25 mg twice daily (bid) for 14 days.
  Interventions: Drug: QBM076
- QBM076 Part 1 Cohort 2 (Experimental): Participants received QBM076 75 mg bid for 14 days.
  Interventions: Drug: QBM076
- QBM076 Part 1 Cohort 3 (Experimental): Participants received QBM076 150 mg bid for 14 days.
  Interventions: Drug: QBM076
- Placebo Part 1 (Placebo Comparator): Participants in each cohort received matching placebo for 14 days.
  Interventions: Drug: Placebo
- QBM076 Part 2 (Experimental): Participants received QBM076 150 mg bid for 8 weeks.
  Interventions: Drug: QBM076
- Placebo Part 2 (Placebo Comparator): Participants received matching placebo for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBM076 — Supplied in 25 mg and 75 mg capsules
  Arms: QBM076 Part 1 Cohort 1; QBM076 Part 1 Cohort 2; QBM076 Part 1 Cohort 3; QBM076 Part 2
Drug: Placebo — Matching placebo capsules
  Other Names: Matching placebo capsules
  Arms: Placebo Part 1; Placebo Part 2

SUMMARY:
This was a 2 Part study. Part 1 was a safety and tolerability study in GOLD I-III COPD patients. Part 2 was an efficacy study in GOLD I-III COPD patients.

DETAILED DESCRIPTION:
Part 1 was a double-blind, randomized, placebo-controlled, non-confirmatory study in chronic bronchitis COPD patients. Part 1 consisted of up to 27-days of screening period, one baseline period of 1 day, 13 days of bid dosing with study treatment, morning only treatment on Day 14, follow up visits on Days 15 - 17, followed by a Study Completion evaluation. Twenty-seven patients were randomized in a 3:1 ratio to 3 cohorts..

Part 2 was a double-blind, randomized, placebo-controlled, non-confirmatory study in Gold spirometry grades I-III COPD patients. Part 2 consisted of up to 20 days of screening period, a 9 day run in period, one baseline period of 1 day, 55 days of bid dosing, morning only dosing on Day 56, followed by Study Completion evaluation. It was planned to randomize 90 patients in a 2:1 ratio, but part 2 was terminated after 21 patients were enrolled. Three of the 21 part 2 patients experienced moderate to severe (up to 17-fold) asymptomatic and reversible elevation of liver transaminase levels after 3 weeks of treatment with QBM076 150 mg twice daily. Two of these patients had liver transaminase levels high enough to be reported as serious adverse events suspected to be related to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Patients, smokers or ex-smokers with stable chronic bronchitis GOLD class I-III chronic obstructive pulmonary disease (COPD); forced expiratory volume in 1 second ≥40% of predicted and forced expiratory volume in 1 second:forced vital capacity ratio ≤0.7 post bronchodilator, respectively; diffusing capacity of the lung for carbon monoxide ≥40%; a stable medical regimen for at least 4 weeks prior to screening. Current smokers can be enrolled if they currently smoke ≤1ppd for last 3 months.

  * Part 2: Patients, smokers or ex-smokers with GOLD spirometry class I-III COPD; a stable medical regimen for at least 4 weeks prior to screening; high sensitivity C reactive protein≥1.5 mg/L; forced expiratory volume in 1 second ≥30% of predicted and forced expiratory volume in 1 second:forced vital capacity ratio ≤0.7 post bronchodilator, respectively; with mean lung clearance index 2.5% ≥8; Ex-smokers with at least 10 pack year smoking history; or current smokers with at least 10 pack year smoking history who smoke ≤ 1ppd on average for last 3 months.; evidence of air trapping based on radiologic criteria; women of child bearing potential using effective methods of contraception

Exclusion Criteria:

* Part 1:Gold Class IV COPD, of moderate to significant emphysema, or evidence of malignancy; medication considered potential for drug drug interaction; creatinine clearance <30ml/min; more than 1 exacerbation requiring antibiotics or oral steroids and/or hospitalization within 3 months of screening; women of child bearing potential • Part 2: Gold spirometry grade IV COPD; medication considered a potential for drug drug interaction; serum creatinine ≥1.9 mg/dL; more than 1 exacerbation requiring antibiotics or oral steroids within 2 months and/or hospitalization within 3 months of screening; any malignancy; evidence of severe emphysema as determined by HRCT; use of oral steroids, theophylline, phosphodiesterase-4 inhibitors or oral antibiotic use (eg.macrolides)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Richmond, Virginia, United States
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In part 1, participants were randomly assigned to one of two treatment arms in a ratio of 3:1 for each cohort. In part 2, participants were stratified by smoking status (current versus ex-smoker) and randomized in a ratio of 2:1 into one of two treatments.
Groups:
- QBM076 Part 1 Cohort 1: Participants received QBM076 25 mg bid for 14 days.
- Placebo Part 1: Participants in each cohort received matching placebo bid for 14 days.
- Placebo Part 2: Participants received matching placebo bid for 8 weeks.
Period: Part 1
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1 | QBM076 Part 2 | Placebo Part 2
Started | 6 | 6 | 8 | 7 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0
Period: Part 2
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1 | QBM076 Part 2 | Placebo Part 2
Started | 0 | 0 | 0 | 0 | 14 | 7
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 13 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1 | QBM076 Part 2 | Placebo Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 14 | 7 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (5.6) | 64 (7.5) | 65 (4.5) | 61 (2.9) | 64 (5.5) | 66 (5.6) | 64 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 4 | 7 | 5 | 24
  Male | 4 | 4 | 4 | 3 | 7 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (Part 1)
Description: Adverse events were counted and corresponding percentages were tabulated.
Time Frame: 14 days
Population: All randomized part 1 participants
Measure: Number; unit: percentage of participants
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1
Number analyzed (Participants) | 6 | 6 | 8 | 7
percentage of participants | 33 | 50 | 63 | 71

2. Primary Outcome: Change From Baseline in Lung Clearance Index (LCI) (Part 2)
Time Frame: Baseline, 8 weeks
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline in Absolute Number of Sputum Neutrophils (Part 2)
Time Frame: Baseline, 8 weeks
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline in Transition Dyspnea Index (TDI) (Part 2)
Time Frame: Baseline, 8 weeks
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) (Part 2)
Time Frame: Baseline, 8 weeks
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval, Tau (AUCtau) (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 1 (from pre-dose to 12 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
ng*h/mL | 431 (158) | 2060 (829) | 7640 (6770)

7. Secondary Outcome: AUCtau, Steady State (AUCtau,ss) (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 14 (from pre-dose to 72 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
ng*h/mL | 601 (112) | 2220 (787) | 6660 (4320)

8. Secondary Outcome: Observed Maximum Plasma Concentration Following Drug Administration (Cmax) (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 1 (from pre-dose to 12 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
ng/mL | 69.5 (28.8) | 366 (192) | 1810 (1790)

9. Secondary Outcome: Cmax,ss (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 14 (from pre-dose to 72 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
ng/mL | 91.0 (13.9) | 338 (123) | 2380 (2680)

10. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 1 (from pre-dose to 12 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Median (Full Range); unit: hours
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
hours | 3.05 [2.00 to 6.00] | 3.01 [2.00 to 8.00] | 3.04 [2.02 to 10.1]

11. Secondary Outcome: Tmax,ss (Part 1)
Description: Venous blood samples were collected for concentration-time profiles.
Time Frame: day 14 (from pre-dose to 72 hours post dose)
Population: All Part 1 participants who received active treatment.
Measure: Median (Full Range); unit: hours
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3
Number analyzed (Participants) | 6 | 6 | 8
hours | 2.00 [2.00 to 4.00] | 2.00 [2.00 to 6.02] | 2.05 [0.50 to 6.02]

12. Secondary Outcome: Change From Baseline in Cluster of Differentiation 11b (CD11b) (Part 1)
Description: Whole blood samples were taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein in order to measure CD11b expression on neutrophils. A negative change from baseline indicates improvement.
Time Frame: baseline, day 14
Population: All Randomized Part 1 participants were considered for the analysis but participants with both baseline and day 14 values were analyzed.
Measure: Number; unit: percentage change
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 5
percentage change | -69 | -89 | -75 | -37

13. Secondary Outcome: Change From Baseline in Chemokine (C-X-C Motif) Receptor 2 (CXCR2) Receptor Occupancy (Part 1)
Description: Whole blood samples were taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein in order to measure CXCR2 receptor occupancy on neutrophils. A positive change from baseline indicates improvement.
Time Frame: baseline, day 14
Population: as for outcome 12
Measure: Number; unit: percent change
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6
percent change | 98 | 104 | 129 | 37

14. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) (Part 1)
Description: FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry and performed at approximately the same time of day on each visit to avoid diurnal variation. All spirometry calibrations and evaluations followed the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability. A positive change from baseline in FEV1 indicates improvement in lung function.
Time Frame: baseline, day 14 pre-dose
Population: as for outcome 12
Measure: Mean (Standard Error); unit: mL
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL | -0.116 (0.05) | -0.008 (0.05) | 0.117 (0.05) | 0.039 (0.05)

15. Secondary Outcome: Change From Baseline in Lung Clearance Index 2.5 (LCI2.5) (Part 1)
Description: Lung clearance index (LCI) is a measure of abnormal ventilation distribution derived from the multiple breath inert gas washout (MBW) technique. LCI is equal to the cumulative expired volume/functional residual capacity. LCI was measured at baseline and day 14. LCI was analyzed using a Bayesian model for repeated measurements. The model may investigate effects for pre-dose baseline, treatment, time, age, COPD class, treatment by time interaction, and baseline by time interaction. A positive change from baseline indicates improvement.
Time Frame: baseline, day 14 pre-dose
Population: as for outcome 12
Measure: Mean (Standard Error); unit: index score
Arm/Group | QBM076 Part 1 Cohort 1 | QBM076 Part 1 Cohort 2 | QBM076 Part 1 Cohort 3 | Placebo Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6
index score | 1.145 (0.42) | 0.136 (0.42) | 0.660 (0.42) | 0.063 (0.42)

16. Secondary Outcome: Change From Baseline in Forced Expirtory Flow 25-75 (FEF25-75), Forced Expiratory Volume 3 (FEV3)/Forced Vital Capacity (FVC), 1-(FEV3/FVC), FEV6, FEV1/FEV6 and Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) (Part 2)
Time Frame: baseline, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: AUC0-24 (Part 2)
Time Frame: day 1, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cmax Between 0h and 24h (Part 2)
Time Frame: day 1, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Tmax Between 0h and 24h (Part 2)
Time Frame: day 1, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Percentage Sputum Neutrophils (Part 2)
Time Frame: baseline, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLco) (Part 2)
Time Frame: baseline, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Scond/Sacin as Measured by Multiple Breath Nitrogen Washout (MBNW) (Part 2)
Time Frame: baseline, day 56
Population: Part 2 was terminated early. Therefore, primary and secondary outcomes for part 2 were not assessed.
Arm/Group | QBM076 Part 2 | Placebo Part 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Part 1: QBM076 B.I.D 25 mg: Part 1: QBM076 B.I.D 25 mg
- Part 1: QBM076 B.I.D 75 mg: Part 1: QBM076 B.I.D 75 mg
- Part 1: QBM076 B.I.D 150 mg: Part 1: QBM076 B.I.D 150 mg
- Part 1: Placebo: Part 1: Placebo
- Part 2: QBM076 B.I.D 150 mg: Part 2: QBM076 B.I.D 150 mg
- Part 2:QBM076 B.I.D Placebo: Part 2:QBM076 B.I.D Placebo
Arm/Group | Part 1: QBM076 B.I.D 25 mg | Part 1: QBM076 B.I.D 75 mg | Part 1: QBM076 B.I.D 150 mg | Part 1: Placebo | Part 2: QBM076 B.I.D 150 mg | Part 2:QBM076 B.I.D Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 1/7 | 2/14 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 5/8 | 4/7 | 8/14 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: QBM076 B.I.D 25 mg (N=6) | Part 1: QBM076 B.I.D 75 mg (N=6) | Part 1: QBM076 B.I.D 150 mg (N=8) | Part 1: Placebo (N=7) | Part 2: QBM076 B.I.D 150 mg (N=14) | Part 2:QBM076 B.I.D Placebo (N=7)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: QBM076 B.I.D 25 mg (N=6) | Part 1: QBM076 B.I.D 75 mg (N=6) | Part 1: QBM076 B.I.D 150 mg (N=8) | Part 1: Placebo (N=7) | Part 2: QBM076 B.I.D 150 mg (N=14) | Part 2:QBM076 B.I.D Placebo (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Catheter site eczema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Therapeutic response unexpected (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Part 2 was terminated after 21 patients were enrolled. Three of the 21 patients experienced moderate to severe (up to 17-fold) asymptomatic and reversible elevation of liver transaminase levels after 3 weeks of treatment with QBM076 150 mg bid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.